CLINICAL TRIAL: NCT06308861
Title: A Dose Block-randomized, Double-blind, Placebo Controlled, Single and Multiple-dosing, Dose-escalation Phase 1 Clinical Trial to Investigate the Safety, Tolerability, PK/PD of J2H-1702 After Oral Administration in Healthy Male Subjects
Brief Title: Investigate Safety, Tolerability, PK/PK of J2H 1702 in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: J2H Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JH-201-101
Record Dates: First submitted 2024-03-05; First posted 2024-03-13 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-02

CONDITIONS: Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (20):
- Single administration Amg dose Group (Experimental)
  Interventions: Drug: Single administration Amg dose Group
- Single administration Bmg dose Group (Experimental)
  Interventions: Drug: Single administration Bmg dose Group
- Single administration Cmg dose Group (Experimental)
  Interventions: Drug: Single administration Cmg dose Group
- Single administration Dmg dose Group (Experimental)
  Interventions: Drug: Single administration Dmg dose Group
- Single administration Emg dose Group (Experimental)
  Interventions: Drug: Single administration Emg dose Group
- Single administration Amg dose Group-Placebo (Placebo Comparator)
  Interventions: Drug: Single administration Amg dose Group-Placebo
- Single administration Bmg dose Group-Placebo (Placebo Comparator)
  Interventions: Drug: Single administration Bmg dose Group-Placebo
- Single administration Cmg dose Group-Placebo (Placebo Comparator)
  Interventions: Drug: Single administration Cmg dose Group-Placebo
- Single administration Dmg dose Group-Placebo (Placebo Comparator)
  Interventions: Drug: Single administration Dmg dose Group-Placebo
- Single administration Emg dose Group-Placebo (Placebo Comparator)
  Interventions: Drug: Single administration Emg dose Group-Placebo
- Multiple administration Amg dose group (Experimental)
  Interventions: Drug: Multiple administration Amg dose group
- Multiple administration Bmg dose group (Experimental)
  Interventions: Drug: Multiple administration Bmg dose group
- Multiple administration Cmg dose group (Experimental)
  Interventions: Drug: Multiple administration Cmg dose group
- Multiple administration Dmg dose group (Experimental)
  Interventions: Drug: Multiple administration Dmg dose group
- Multiple administration Emg dose group (Experimental)
  Interventions: Drug: Multiple administration Emg dose group
- Multiple administration Amg dose group - Placebo (Placebo Comparator)
  Interventions: Drug: Multiple administration Amg dose group - Placebo
- Multiple administration Bmg dose group - Placebo (Placebo Comparator)
  Interventions: Drug: Multiple administration Bmg dose group - Placebo
- Multiple administration Cmg dose group - Placebo (Placebo Comparator)
  Interventions: Drug: Multiple administration Cmg dose group - Placebo
- Multiple administration Dmg dose group - Placebo (Placebo Comparator)
  Interventions: Drug: Multiple administration Dmg dose group - Placebo
- Multiple administration Emg dose group - Placebo (Placebo Comparator)
  Interventions: Drug: Multiple administration Emg dose group - Placebo

INTERVENTIONS:
Drug: Single administration Amg dose Group — Orally, Amg tablet single administration
  Arms: Single administration Amg dose Group
Drug: Single administration Bmg dose Group — Orally, Bmg tablet single administration
  Arms: Single administration Bmg dose Group
Drug: Single administration Cmg dose Group — Orally, Cmg tablet single administration
  Arms: Single administration Cmg dose Group
Drug: Single administration Dmg dose Group — Orally, Dmg tablet single administration
  Arms: Single administration Dmg dose Group
Drug: Single administration Emg dose Group — Orally, Emg tablet single administration
  Arms: Single administration Emg dose Group
Drug: Single administration Amg dose Group-Placebo — Orally, Placebo Amg tablet, single administration
  Arms: Single administration Amg dose Group-Placebo
Drug: Single administration Bmg dose Group-Placebo — Orally, Placebo Bmg tablet, single administration
  Arms: Single administration Bmg dose Group-Placebo
Drug: Single administration Cmg dose Group-Placebo — Orally, Placebo Cmg tablet, single administration
  Arms: Single administration Cmg dose Group-Placebo
Drug: Single administration Dmg dose Group-Placebo — Orally, Placebo Dmg tablet, single administration
  Arms: Single administration Dmg dose Group-Placebo
Drug: Single administration Emg dose Group-Placebo — Orally, Placebo Emg tablet, single administration
  Arms: Single administration Emg dose Group-Placebo
Drug: Multiple administration Amg dose group — Orally, Amg 1 tablet, once a day for 3 days, multiple administration
  Arms: Multiple administration Amg dose group
Drug: Multiple administration Bmg dose group — Orally, Bmg 1 tablet, once a day for 3 days, multiple administration
  Arms: Multiple administration Bmg dose group
Drug: Multiple administration Cmg dose group — Orally, Cmg 1 tablet, once a day for 3 days, multiple administration
  Arms: Multiple administration Cmg dose group
Drug: Multiple administration Dmg dose group — Orally, Dmg 1 tablet, once a day for 3 days, multiple administration
  Arms: Multiple administration Dmg dose group
Drug: Multiple administration Emg dose group — Orally, Emg 1 tablet, once a day for 3 days, multiple administration
  Arms: Multiple administration Emg dose group
Drug: Multiple administration Amg dose group - Placebo — Orally, Placebo Amg 1 tablet, once a day for 3 days, multiple administration
  Arms: Multiple administration Amg dose group - Placebo
Drug: Multiple administration Bmg dose group - Placebo — Orally, Placebo Bmg 1 tablet, once a day for 3 days, multiple administration
  Arms: Multiple administration Bmg dose group - Placebo
Drug: Multiple administration Cmg dose group - Placebo — Orally, Placebo Cmg 1 tablet, once a day for 3 days, multiple administration
  Arms: Multiple administration Cmg dose group - Placebo
Drug: Multiple administration Dmg dose group - Placebo — Orally, Placebo Dmg 1 tablet, once a day for 3 days, multiple administration
  Arms: Multiple administration Dmg dose group - Placebo
Drug: Multiple administration Emg dose group - Placebo — Orally, Placebo Emg 1 tablet, once a day for 3 days, multiple administration
  Arms: Multiple administration Emg dose group - Placebo

SUMMARY:
1. Research Purpose: To evaluate the safety, tolerability, pharmacokinetic/pharmacodynamic properties of J2H-1702 (a candidate for treatment of non-alcoholic steatohepatitis) in healthy men.
2. Design: A dose block-randomized, double-blind, placebo controlled, single- and multiple dosing, dose-escalation phase 1 clinical trial

DETAILED DESCRIPTION:
Subjects in all dose groups will be randomized to the study group (J2H-1702 group) and the control group (Placebo group) in a 8:2 ratio. Adverse event (AE) collection, physical examination, vital signs, ECG, clinical laboratory tests, etc. will be performed to assess the safety and tolerability, and blood and urine sampling will be performed to assess the PK/PD characteristics. In addition, blood sampling for mass cytometry (multiple administration study) and baseline fibroscan will be performed for the exploratory evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. A healthy male adult within the range of 19 to 45 years old
2. BMI=18.0~27.0kg/m2 (Body mass index, BMI)
3. A subject confirmed to be clinically healthy based on the medical history, physical examination, vitals signs, ECG, and appropriate clinical laboratory tests
4. A subject who his spouse or partner agrees to use dual contraceptive methods and not to donate sperms
5. A subject who has voluntarily agree to participate in the study

Exclusion Criteria:

1. A subject who had or has the disease corresponding to clinically significant liver, etc.
2. A subject with a history of gastrointestinal diseases or surgery
3. A subject who has a history of clinically significant hypersensitivity to drugs containing 11β-HSD1 inhibitor
4. A subject who has genetic problems such as galactose intolerance, Lap galactose intolerance, Lap lactase deficiencies, or glucose ∙galactose malabsorptivity, etc.
5. One who has drug abuse and one who is positive response in urine drug screening tests
6. A subject with abnormal vital signs at the screening visit
7. A subject who has participated in another clinical trial or bioequivalence test
8. A subject who donated whole blood or the ingredient, or received blood transfusion
9. A subject who took drug metabolizing enzyme-inducing and inhibitory drugs
10. A subject who consumes grapefruit/caffeine-containing food
11. A subject who took any prescription drug or herbal medicine or took any Over The Counter Drug (OTC)
12. High caffeine intaker, high alcohol intaker or excessive smoker
13. A subject who cannot eat meals provided by the Clinical Trial institution.
14. A subject who participated in this trial and were administered the investigational product.
15. A subject who is positive for serum test
16. A subject who the investigator deems inappropriate for this clinical trial.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Cmax | 1day 0 (Before IP administration), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36, 48 hours (After IP administration)
  Pharmacokinetics
Emax | -1day 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 hours, 1day 0 (Before IP administration), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24hours (After IP administration)
  Pharmacodynamics

CONTACTS AND LOCATIONS:
Locations (1):
- J2H Biotech, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No